CLINICAL TRIAL: NCT01098526
Title: A Phase 1, Open Label, Single Sequence, Three Period Study to Evaluate the Single Dose Pharmacokinetics of GSK1349572 100mg Versus 50mg and the Effect of Efavirenz 600mg Once Daily on the Pharmacokinetics, Safety and Tolerability of GSK1349572 50mg Once Daily in Healthy Adult Subjects (ING114005)
Brief Title: GSK1349572 Drug Interaction Study With Efavirenz
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: ViiV Healthcare (Industry)
Collaborators: Shionogi (Industry); GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 114005
Record Dates: First submitted 2010-03-04; First posted 2010-04-02 (Estimated); Last update posted 2017-09-25 (Actual); Status verified 2017-09

CONDITIONS: Infections, Human Immunodeficiency Virus and Herpesviridae
Keywords: GSK1349572; efavirenz; integrase; pharmacokinetics
MeSH Terms: conditions — Infections; Acquired Immunodeficiency Syndrome | interventions — dolutegravir; efavirenz

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Cohort 1 (Experimental): Subjects will receive a single dose of GSK1349572 100 mg in Period 1 followed by a washout of at least 6 days. Subjects will then receive GSK1349572 50 mg once a day for 5 days in Period 2. Period 3 will begin immediately after Period 2. In Period 3 subjects will receive GSK1349572 50 mg once a day in the morning and Efavirenz 600 mg once a day at bedtime for 14 days. There will be a screening visit up to 30 days before Period 1 and a follow up visit 7-14 days after the end of Period 3.
  Interventions: Drug: GSK1349572; Drug: Efavirenz

INTERVENTIONS:
Drug: GSK1349572 — GSK1349572 is an experimental drug under development for the treatment of HIV. It is in the class of integrase inhibitors.
Drug: Efavirenz — Efavirenz is a drug that has been approved by the FDA for the treatment of HIV. It is in the class of non-nucleoside reverse trancriptase inhibitors.
  Other Names: SUSTIVA. SUSTIVA is a registered trademark of Bristol-Myers Squibb

SUMMARY:
GSK1349572 is an integrase inhibitor that is currently in Phase 2 clinical trials for the treatment of HIV infection. As GSK1349572 development progresses, it may be dosed with non-nucleoside HIV reverse transcriptase inhibitors (NNRTIs) including efavirenz (EFV, Sustiva). Efavirenz is a known inducer of CYP3A4. GSK1349572 is primarily metabolized via UGT1A1, however it also has a CYP component to its metabolism, thus a drug interaction between GSK1349572 and EFV is likely. A previous study showed that another NNRTI, etravirine which is also a known inducer of CYP3A and UGT, reduced GSK1349572 exposure significantly. GSK1349572 is not an inhibitor or inducer of CYP3A and is not expected to have impact on pharmacokinetics (PK) of EFV.

This study will investigate the dose proportionality between single doses of 50mg and 100mg of GSK1349572 and will compare steady-state plasma PK, safety and tolerability of GSK1349572 50 mg every 24h (q24h) with and without efavirenz 600 mg q24h. Approximately 12 subjects will receive a single dose of GSK1349572 100 mg (Treatment A) in Period 1 followed by a washout of greater than or equal to 6 days. In Period 2 subjects will receive GSK1349572 50mg q24h for 5 days (Treatment B). Subjects will then be administered GSK1349572 50mg q24h in the morning in combination with EFV 600 mg q24h (Treatment C) in the evening for 14 days in Period 3. There will be no washout between Periods 2 and 3. Safety evaluations and serial PK samples for GSK1349572 will be collected during each treatment period. A follow-up visit will occur 7-14 days after the last dose of study drug.

This study will be conducted at one center in the US, with healthy adult male and female subjects.

DETAILED DESCRIPTION:
ViiV Healthcare is the new sponsor of this study, and GlaxoSmithKline is in the process of updating systems to reflect the change in sponsorship.

ELIGIBILITY:
Inclusion Criteria:

* AST, ALT, alkaline phosphatase and bilirubin less than or equal to 1.5xULN (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35%).
* Healthy as determined by a responsible and experienced physician, based on a medical evaluation including medical history, physical examination, laboratory tests and cardiac monitoring.
* Male or female between 18 and 65 years of age inclusive, at the time of signing the informed consent.
* A female subject is eligible to participate if she is of: Non-childbearing potential defined as pre-menopausal females with a documented tubal ligation or hysterectomy; or postmenopausal defined as 12 months of spontaneous amenorrhea [in questionable cases a blood sample with simultaneous follicle stimulating hormone (FSH) > 40 MlU/ml and estradiol < 40 pg/ml (<147 pmol/L) is confirmatory].
* Body weight greater than or equal to 50 kg for males and 45 kg for females and BMI within the range 18.5- 31.0 kg/m2 (inclusive).
* Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form.

Exclusion Criteria:

* The subject has a positive pre-study drug/alcohol screen. A minimum list of drugs that will be screened for include amphetamines, barbiturates, cocaine, opiates, cannabinoids and benzodiazepines.
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
* History of sensitivity to any of the study medications, or components thereof, or a history of drug or other allergy that, in the opinion of the investigator or GSK Medical Monitor, contraindicates their participation.
* Use of prescription or non-prescription drugs, including vitamins, herbal and dietary supplements (including St John's Wort) within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to the first dose of study medication, unless in the opinion of the Investigator and GSK Medical Monitor the medication will not interfere with the study procedures or compromise subject safety.
* If heparin is used during PK sampling, subjects with a history of sensitivity to heparin or heparin-induced thrombocytopenia should not be enrolled.
* History of regular alcohol consumption within 6 months of the study defined as an average weekly intake of >14 drinks/week for men or >7 drinks/week for women. One drink is equivalent to (12 g alcohol) = 5 ounces (150 ml) of wine or 12 ounces (360 ml) of beer or 1.5 ounces (45 ml) of 80 proof distilled spirits.
* Has a history or regular use of tobacco- or nicotine-containing products within 3 months prior to screening.
* Consumption of red wine, seville oranges, grapefruit or grapefruit juice from 7 days prior to the first dose of study medication.
* Pregnant females as determined by positive serum or urine human chorionic gonadotrophin (hCG) test at screening or prior to dosing.
* Lactating females.
* Unwillingness or inability to follow the procedures outlined in the protocol.
* Subjects with a pre-existing condition interfering with normal gastrointestinal anatomy or motility, hepatic and/or renal function, that could interfere with the absorption, metabolism, and/or excretion of the study drugs. Subjects with a history of cholecystectomy, peptic ulceration, inflammatory bowel disease or pancreatitis should be excluded.
* History/evidence of symptomatic arrhythmia, angina/ischemia, coronary artery bypass grafting (CABG) surgery or percutaneous transluminal coronary angioplasty (PCTA) or any clinically significant cardiac disease.
* History/evidence of clinically significant pulmonary disease.
* History of significant renal or hepatobiliary diseases. Subjects with a history of nephrolithiasis will be excluded.
* History of severe or serious psychiatric disease ever requiring hospitalization, history of suicidal ideation or suicidal attempt, or undergoing psychiatric treatment will be excluded from study participation.
* A positive pre-study Hepatitis B surface antigen or positive Hepatitis C antibody result within 3 months of screening.
* A positive test for HIV antibody.
* History of 2nd degree or higher AV block.
* History of Gilbert's disease.
* Where participation in the study would result in donation of blood or blood products in excess of 500 mL within a 56 day period.
* The subject's systolic blood pressure is outside the range of 90-140mmHg, or diastolic blood pressure is outside the range of 45-90mmHg or heart rate is outside the range of 50-100bpm for female subjects or 45-100 bpm for male subjects.
* Exclusion criteria for screening ECG per protocol

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2010-03-16 (Actual); Primary Completion 2010-05-26 (Actual); Study Completion 2010-05-26 (Actual)

PRIMARY OUTCOMES:
Plasma GSK1349572 PK parameters: AUC (0-24) | 24 hours
  Plasma GSK1349572 PK parameters: AUC(0-24), Cmax, and C24, and dose-normalized AUC(0-24), Cmax, and C24 following single dose administration of 100mg and 50mg.
Plasma GSK1349572 PK parameters: Cmax | 24 hours
  Plasma GSK1349572 PK parameters: AUC(0-24), Cmax, and C24, and dose-normalized AUC(0-24), Cmax, and C24 following single dose administration of 100mg and 50mg.
Plasma GSK1349572 PK parameters: C24 | 24 hours
  Plasma GSK1349572 PK parameters: AUC(0-24), Cmax, and C24, and dose-normalized AUC(0-24), Cmax, and C24 following single dose administration of 100mg and 50mg.
Plasma GSK1349572 steady-state AUC (0-tau) | 19 days
  Plasma GSK1349572 steady-state AUC(0-tau), Cmax, C0, Ctau, and Cmin following administration of GSK1349572 50mg q24h for 5 days and following co-administration with EFV 600mg q24h for 14 days.
Plasma GSK1349572 steady-state Cmax | 19 days
  Plasma GSK1349572 steady-state AUC(0-tau), Cmax, C0, Ctau, and Cmin following administration of GSK1349572 50mg q24h for 5 days and following co-administration with EFV 600mg q24h for 14 days.
Plasma GSK1349572 steady-state C0 | 19 days
  Plasma GSK1349572 steady-state AUC(0-tau), Cmax, C0, Ctau, and Cmin following administration of GSK1349572 50mg q24h for 5 days and following co-administration with EFV 600mg q24h for 14 days.
Plasma GSK1349572 steady-state Ctau | 19 days
  Plasma GSK1349572 steady-state AUC(0-tau), Cmax, C0, Ctau, and Cmin following administration of GSK1349572 50mg q24h for 5 days and following co-administration with EFV 600mg q24h for 14 days.
Plasma GSK1349572 steady-state Cmin | 19 days
  Plasma GSK1349572 steady-state AUC(0-tau), Cmax, C0, Ctau, and Cmin following administration of GSK1349572 50mg q24h for 5 days and following co-administration with EFV 600mg q24h for 14 days.

SECONDARY OUTCOMES:
Safety and tolerability parameters | 4 weeks
  Safety and tolerability parameters, including adverse event, concurrent medication, clinical laboratory, ECG, and vital signs assessments.
Plasma GSK1349572 single dose PK parameters: tmax | 24 hours
  Plasma GSK1349572 single dose PK parameters: tmax and tlag, following administration of GSK1349572 100mg and 50mg.
Plasma GSK1349572 single dose PK parameters: tlag | 24 hours
  Plasma GSK1349572 single dose PK parameters: tmax and tlag, following administration of GSK1349572 100mg and 50mg.
Plasma GSK1349572 steady-state PK parameters: tmax | 19 days
  Plasma GSK1349572 steady-state PK parameters: tmax, tmin, CL/F, and t½, following 50mg q24h for 5 days and following co-administration with EFV 600mg q24h for 14 days.
Plasma GSK1349572 steady-state PK parameters: tmin | 19 days
  Plasma GSK1349572 steady-state PK parameters: tmax, tmin, CL/F, and t½, following 50mg q24h for 5 days and following co-administration with EFV 600mg q24h for 14 days.
Plasma GSK1349572 steady-state PK parameters: CL/F | 19 days
  Plasma GSK1349572 steady-state PK parameters: tmax, tmin, CL/F, and t½, following 50mg q24h for 5 days and following co-administration with EFV 600mg q24h for 14 days.
Plasma GSK1349572 steady-state PK parameters: t½ | 19 days
  Plasma GSK1349572 steady-state PK parameters: tmax, tmin, CL/F, and t½, following 50mg q24h for 5 days and following co-administration with EFV 600mg q24h for 14 days.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — ViiV Healthcare
Locations (1):
- GSK Investigational Site, Buffalo, New York, United States